CLINICAL TRIAL: NCT05754372
Title: Optimalisation of the Treatment of Acute Neonatal Hyperammonaemia
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-10637
Record Dates: First submitted 2022-01-03; First posted 2023-03-03 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Hyperammonemic Encephalopathy
Keywords: hemodialysis; neonate; Hyperammonemic Encephalopathy; inborn error of metbolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma, urine, dialysate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hyperammonaemia
  Interventions: Diagnostic Test: user-friendly and widely applicable algorithm to tailor the treatment of acute neonatal hyperammonemia

INTERVENTIONS:
Diagnostic Test: user-friendly and widely applicable algorithm to tailor the treatment of acute neonatal hyperammonemia — user-friendly and widely applicable algorithm to tailor the treatment of acute neonatal hyperammonemia, based on kinetic modelling

SUMMARY:
Acute neonatal hyperammonemia is associated with poor neurological outcomes and high mortality. A user-friendly and widely applicable algorithm - based on kinetics - to tailor the treatment of acute neonatal hyperammonemia. A single compartmental model was calibrated assuming a distribution volume equal to the patient's total body water (V), as calculated using Wells' formula, and dialyzer clearance as derived from the measured ammonia time-concentration curves during 11 dialysis sessions in four patients (3.2 +/- 0.4 kg). Based on these kinetic simulations, dialysis protocols could be derived for clinical use with different body weights, start concentrations, dialysis machines/dialyzers and dialysis settings (e.g., blood flow QB). By a single measurement of ammonia concentration at the dialyzer inlet and outlet, dialyzer clearance (K) can be calculated as K = QB[(Cinlet - Coutlet)/Cinlet]. The time (T) needed to decrease the ammonia concentration from a predialysis start concentration Cstart to a desired target concentration Ctarget is then equal to T = (-V/K)LN(Ctarget/Cstart). By implementing these formulae in a simple spreadsheet, medical staff can draw an institution-specific flowchart for patient-tailored treatment of hyperammonemia.

The aim of this study is to validate these formula with a prospective study.

ELIGIBILITY:
Inclusion Criteria:

* severe acute neonatal hyperammonaemia for which acute hemodialysis is indicated
* inborn error of metabolism
* below 1 year of age

Exclusion Criteria:

* older than 1 year

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infants presenting with acute neonatale hyperammonaemia
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
serum ammonium levels | 1 year
  serum ammonium levels

SECONDARY OUTCOMES:
Removal of treatment sodium benzoate, L-arginine | 1 year
  serum and dialysate concentration (mg/dL) of sodium benzoate and L-arginine

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital - Department of Paediatric Nephrology, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No